CLINICAL TRIAL: NCT04130425
Title: A Comparison Study of Three Standard Elbow Wrist Hand Orthoses to Limit Forearm Rotation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephanie N. Kannas, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-008562
Record Dates: First submitted 2019-10-13; First posted 2019-10-17 (Actual); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy Individuals (Experimental): Subject will be measured for forearm rotation while wearing the custom orthoses Hely & Weber MTC Fracture Brace, thermoplastic orthosis, and delta cast orthosis.
  Interventions: Device: Hely & Weber MTC Fracture Brace; Device: Thermoplastic orthosis; Device: Delta cast orthosis

INTERVENTIONS:
Device: Hely & Weber MTC Fracture Brace — Prefabricated muenster orthosis
Device: Thermoplastic orthosis — Muenster orthosis fabricated out of thermoplastics and secured with Velcro
Device: Delta cast orthosis — Muenster orthosis fabricated out of Delta Cast and secured with Velcro

SUMMARY:
The Researchers are trying to assess which splint limits forearm rotation the best. These splints are commonly used in hand therapy to limit forearm rotation. This data will help hand surgery and hand therapy provide better outcomes.

DETAILED DESCRIPTION:
Common upper extremity injuries often need to heal with no wrist and forearm range of motion. Forearm range of motion includes supination and pronation. Injuries that necessitate limiting forearm range of motion include fracture patterns involving the distal radioulnar joint (DRUJ), proximal radioulnar joint (PRUJ), triangular fibrocartilage complex (TFCC), both bone forearm fractures, ulnar shortening procedures, radial and ulnar osteotomies, DRUJ instability. Long arm orthoses, sugar tong orthoses and muenster style orthoses can all limit forearm rotation.

Past research has indicated common methods of immobilization to include the following: sugar tongs cast/orthosis, muenster cast/orthosis, long arm cast/orthosis/or short arm cast/orthosis, and an antirotation orthosis.

Currently, there are no research studies that compare the amount of forearm rotation in a traditional thermoplastic orthoses to newer materials such as a Delta Cast orthosis, or prefabricated muenster orthoses such as the Hely and Weber MTC Fracture Brace. The purpose of this study is to assess which orthosis-a traditional thermoplastic ulnar based muenster, a delta cast style muenster and the Hely and Weber MTC Fracture Brace-allows for the least amount of supination and pronation in a healthy population in the dominant extremity.

The researchers will assess the 3 different orthoses using a standard measuring device for pronation and supination. The participants will also be asked questions regarding comfort, fit, and style of each orthosis. 30 Participants data will be collected during the study.

ELIGIBILITY:
Inclusion Criteria:

* No prior wrist or elbow injuries on the dominant side of his/her body
* Ability to complete study in one sitting of 90-120 minutes
* Between the ages of 18 years and 100 years
* Ability to follow directions and speak and read English

Exclusion Criteria:

* Prior wrist or elbow injuries on the dominant side of his/her body
* Subjects with known rheumatoid arthritis deformities of the wrist or any prior wrist surgeries are excluded

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stepanie Kannas, CHT, OT, OTD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Hely & Weber MTC Fracture Brace, Thermoplastic Orthosis and Delta-Cast Orthosis: Each participant received a sequence of three different orthotic interventions and served as his/her own match control to assess forearm range of motion.
Period: Overall Study
Arm/Group | Hely & Weber MTC Fracture Brace, Thermoplastic Orthosis and Delta-Cast Orthosis
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Individuals
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Degree of Forarm Rotation With Thermoplastic Ulnar Based Muenster Orthosis, Delta-Cast Orthosis and Hely and Weber Fracture Brace MTC
Description: Degree of forarm rotation (supination/pronation) measured by an electronic goniometer device reported unit of measurement in degrees while wearing each of the orthoses.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Thermoplastic Results: The 30 healthy participants trialing the thermoplastic orthosis. Total arc of motion reported.
- Delta-Cast Results: The 30 healthy participants trialing the Delta-Cast orthosis. Results are total arc of motion.
- Hely and Weber Fracture Brace MTC: The 30 healthy participants trialing the Hely and Weber Fracture Brace MTC. Results reported in total arc of motion.
Arm/Group | Thermoplastic Results | Delta-Cast Results | Hely and Weber Fracture Brace MTC
Number analyzed (Participants) | 30 | 30 | 30
degrees | 88.4 (35.8) | 49.1 (24.2) | 67.2 (34.5)

2. Secondary Outcome: Orthotics and Prosthetics User's Survey (OPUS )
Description: The OPUS is a well validated, self-report questionnaire which consists of five modules; specifically, five questions from the OPUS: Satisfaction with Device and Services Module were used. These five questions were scored on a 5-point Likert scale from strongly agree to strongly disagree. A sixth option of "don't know" or "not applicable" was also available. Strongly agree = 5, Agree = 4, Neutral =3, Disagree =2, Strongly Disagree =1. If the participant chose don't know or not applicable that question was excluded for that participant.
  The five questions included-
  1. . My orthosis fits well.
  2. . The weight of my orthosis is manageable.
  3. . It is easy to put on my orthosis.
  4. . My orthosis is pain free to wear.
  5. . My orthosis looks good.
  The remaining 16 questions from the module were excluded, as they did not pertain to healthy volunteers wearing the orthosis only during his/her research participation.
Time Frame: 1 day
Population: Participants were excluded from overall analysis if they answered don't know or not applicable for certain questions in the study.
Measure: Mean (Standard Deviation); unit: Likert scale unit
Groups:
- Hely & Weber MTC Fracture Brace: Each participant is their own matched control for the three orthoses. This data describes only the Hely & Weber MTC Fracture Brace.
- Thermoplastic Orthosis: Each participant is their own matched control for the three orthoses. This data describes only the Thermoplastic Orthosis
- Delta-Cast Orthosis: Each participant is their own matched control for the three orthoses. This data describes only the Delta Cast orthosis
Arm/Group | Hely & Weber MTC Fracture Brace | Thermoplastic Orthosis | Delta-Cast Orthosis
Number analyzed (Participants) | 30 | 30 | 30
Likert scale unit
  My orthosis fits well | 4.2 (0.9) | 4.0 (0.7) | 4.7 (0.5)
  The weight is manageable | 4.1 (0.9) | 4.3 (0.7) | 4.4 (0.8)
  Easy to put on orthosis | 3.5 (1.2) | 4.2 (0.8) | 3.8 (1.2)
  My orthosis is pain free to wear: number analyzed (Participants) | 29 | 29 | 29
  My orthosis is pain free to wear | 4.2 (0.9) | 4.0 (0.9) | 4.5 (0.9)
  My orthosis looks good: number analyzed (Participants) | 28 | 28 | 28
  My orthosis looks good | 3.5 (1.2) | 4.2 (0.8) | 3.4 (1.2)

ADVERSE EVENTS:
Time Frame: 1 day
Description: The nature of the study was completing normal standard of care for orthotic positioning. All safety practices were in place that are followed for standard clinic operations.
Groups:
- Hely & Weber MTC Fracture Brace; Thermoplastic Orthosis; Delta-Cast Orthosis: Participants served as their own matched controls for each of the three orthoses.
Arm/Group | Hely & Weber MTC Fracture Brace | Thermoplastic Orthosis | Delta-Cast Orthosis
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
All measurements were performed on healthy individuals versus an injured arm. Since participants did not have symptoms, it made donning and doffing the orthoses easier. During testing, participants were asked to pronate and supinate until they felt resistance using sensory feedback as the stop point. This limitation allowed for the wide variant in allowable motion of each orthosis, as each participant's perception could be different when it comes to feeling resistance in an orthosis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT04130425/Prot_SAP_001.pdf